CLINICAL TRIAL: NCT07118527
Title: A Phase III, Randomized, Multicenter, Open-label Study to Evaluate SHR-A1811 in Combination With Chemotherapy and Adebrelimab Versus Trastuzumab in Combination With Chemotherapy and Pembrolizumab in Patients With Previously Untreated, Unresectable, Locally Advanced or Metastatic, Gastric or Gastroesophageal Junction Adenocarcinoma Expressing
Brief Title: A Phase III Study of SHR-A1811 in Combination With Chemotherapy and Adebrelimab in Previously Untreated Patients With Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-316
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Patients With Unresectable Locally Advanced or Metastatic Untreated Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Capecitabine; Trastuzumab; pembrolizumab; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: (Experimental): SHR-A1811 + Adebrelimab Injection + Capecitabine Tablets or Fluorouracil Injection
  Interventions: Drug: SHR-A1811 + Adebrelimab Injection + Capecitabine Tablets or Fluorouracil Injection
- Treatment group B (Active Comparator): Trastuzumab + Pembrolizumab + CAPOX( Capecitabine Tablets + Oxaliplatin) or FP (Fluorouracil Injection+Cisplatin)
  Interventions: Drug: Trastuzumab + Pembrolizumab + CAPOX( Capecitabine Tablets + Oxaliplatin) or FP (Fluorouracil Injection+Cisplatin)

INTERVENTIONS:
Drug: SHR-A1811 + Adebrelimab Injection + Capecitabine Tablets or Fluorouracil Injection — SHR-A1811: intravenous infusion; Adebrelimab Injection: intravenous infusion; Capecitabine Tablets: oral administration Fluorouracil Injection: intravenous infusion
  Arms: Treatment group A:
Drug: Trastuzumab + Pembrolizumab + CAPOX( Capecitabine Tablets + Oxaliplatin) or FP (Fluorouracil Injection+Cisplatin) — Trastuzumab : intravenous infusion; Pembrolizumab: intravenous infusion; Capecitabine Tablets: oral administration; Oxaliplatin: intravenous infusion; Fluorouracil Injection: intravenous infusion; Cisplatin: intravenous infusion;
  Arms: Treatment group B

SUMMARY:
This study aims to evaluate the efficacy and safety of SHR-A1811 combined with chemotherapy and immune checkpoint inhibitor versus standard first-line therapy in gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years (inclusive), male or female
2. Histologically or cytologically confirmed untreated, locally advanced, unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma.
3. ECOG performance status score of 0 to 1.
4. Body weight ≥ 35 kg.
5. Life expectancy ≥12 weeks.
6. Must have at least one measurable lesion according to RECIST v1.1 criteria.
7. Tumor tissue samples must be provided, and newly obtained tumor tissues are preferred.
8. Adequate bone marrow and organ function；
9. Women of childbearing potential must agree on abstinence (avoid heterosexual sex) or use of the highly effective methods of contraception from the signature of informed consent form until at least 7 months after the last dose of the investigational product(s).
10. Male patients whose partners are women of childbearing potential must agree on abstinence or use of the highly effective methods of contraception from the signature of informed consent form until at least 7 months after the last dose of investigational product(s).
11. Capable of giving informed consent, have signed and dated the informed consent approved by the Ethics Committee, and willing and able to comply with tests and other procedures at scheduled visits.

Exclusion Criteria:

1. Current or previous meningeal metastases; presence of active brain metastases.
2. Ascites, pleural effusion and pericardial effusion requiring treatment (such as puncture, drainage, etc.) within 2 weeks before randomization.
3. Subjects with other malignant tumors within 3 years before randomization.
4. Have received traditional Chinese medicine with anti-tumor indications within 2 weeks before randomization.
5. With adverse reactions (ARs) from previous anti-tumor treatment that have not recovered to NCI-CTCAE v5.0 Grade ≤ 1.
6. Use of other non-marketed clinical investigational products or interventions within 4 weeks before randomization.
7. Have undergone major surgery (excluding aspiration biopsy) or experienced significant trauma within 4 weeks before randomization.
8. Patients with active autoimmune diseases or history of autoimmune diseases.
9. Patients with known or suspected interstitial lung disease; patients with other severe lung diseases that seriously affect respiratory function within 3 months before randomization.
10. History of active tuberculosis within 1 year before randomization, or history of active tuberculosis over 1 year without appropriate treatment.

11、14. History of immunodeficiency, including positive HIV test; active hepatitis B or hepatitis C.

12、Patients who have previously undergone allogeneic hematopoietic stem cell transplantation or organ transplantation.

13、Severe cardiovascular or cerebrovascular diseases. 14、Active bleeding (CTCAE Grade ≥ 2). 15、Gastrointestinal perforation, gastrointestinal fistula or abdominal infection within 3 months before randomization.

16、Uncontrollable tumor-related pain or symptomatic hypercalcemia. 17、Patients with Grade > 1 peripheral neuropathy. 18、Vaccination of live attenuated vaccine within 28 days prior to randomization.

19、Previous use of anti-HER2 antibody-drug conjugates.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per RECIST 1.1 assessed by BIRC(Blinded Independ Review Committee) | UP to approximately 5 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first.
Overall Survival （OS） | UP to approximately 5 years
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 assessed by BIRC | UP to approximately 5 years
  ORR is defined as the proportion of participants who have a complete response (CR) or partial response (PR)
PFS per RECIST 1.1 assessed by investigator | UP to approximately 5 years
  PFS is defined as time from randomization until progression per RECIST v1.1, or death due to any cause.
Disease Control Rate (DCR) per RECIST 1.1 | UP to approximately 5 years
  DCR is defined as the proportion of patients who exhibit no tumor progression (including shrinkage or stability) after treatment.
Duration of Response (DOR) | UP to approximately 5 years
  DOR is defined as the time from the first achievement of complete response (CR) or partial response (PR) to the first occurrence of disease progression (PD) or death from any cause.
Adverse events (AE) | UP to approximately 5 years
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Zhongshan Hospital，Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided